CLINICAL TRIAL: NCT06204744
Title: Scale-out of a Home-based Arm and Hand Exercise Program for Stroke: A Multisite Implementation-efficacy Trial
Brief Title: Home-based Arm and Hand Exercise Program for Stroke: A Multisite Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chieh-ling Yang, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202200321B0
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based GRASP program (Experimental)
  Interventions: Other: Home-based GRASP program
- Conventional occupational therapy home program (Active Comparator)
  Interventions: Other: Conventional occupational therapy home program

INTERVENTIONS:
Other: Home-based GRASP program — The home-based Graded Repetitive Arm Supplementary Program (GRASP) is designed to improve the upper extremity function for people with stroke, including exercises for stretching, coordination, arm and hand strengthening, and fine motor skills.
  Arms: Home-based GRASP program
Other: Conventional occupational therapy home program — The conventional OT home program will be prescribed by the occupational therapists, customizing stroke rehabilitation exercises to individual patient goals, with a primary focus on improving upper extremity function.
  Arms: Conventional occupational therapy home program

SUMMARY:
The goal of this multisite clinal trial is to evaluate the implementation of the home-based Graded Repetitive Arm Supplementary Program (GRASP) at rehabilitation clinics across several hospitals. The main questions it aims to answer is:

• the efficacy of the home-based GRASP program relative to the conventional occupational therapy intervention on improving health outcomes, including UE motor function, daily function, quality of life, and motor control strategies.

Stroke participants will be randomly assigned to either the Home-based GRASP group or the conventional occupational therapy home program group. Each group will undergo an 4 to 6-week intervention (3 sessions/week) with evaluations conducted before, immediately after, and 3 months post-trial, assessing clinical and kinematic measures. Interviews and surveys will be conducted to gain insights into the perspectives of patients regarding the implementation of the home-based GRASP program.

ELIGIBILITY:
Inclusion Criteria:

* are aged 20 years or older
* have upper extremity hemiparesis due to the first-ever stroke
* have some voluntary movement in the affected UE
* are able to follow 2-step instructions

Exclusion criteria:

* orthopedic conditions affecting the arm/hand or other neurological conditions
* severe pain that prevents movement in the affected arm and hand
* unstable medical status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (upper extremity) | Baseline, post-test (1 month after baseline), 3-month followup
  The FMA-UE is one of the most widely used assessments to quantify UE sensorimotor impairment of the shoulder, elbow, forearm, wrist, and hand. It is based on a 3-point scale (0 cannot perform; 1 can perform partially; 2 can perform fully). The total scores range between 0 and 66, with a higher FMA-UE score indicating less motor impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-ling Yang, Principal Investigator — Chang Gung University
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided